CLINICAL TRIAL: NCT05376436
Title: The Effect of Mouth Breathing on Exercise Induced Bronchoconstriction in Children.
Brief Title: Effect of Mouth Breathing on Exercise Induced Bronchoconstriction.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0716-19-RMB
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Asthma in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exercise challenge test (ECT) with and without nose clip (NC).: All participants after receiving informed consent were invited for 2 visits. Visit 1 - ECT performed with NC. Visit 2 - ECT performed without NC. Demographic and clinical data and measurements of vital signs, exercise data and lung functions were recorded.
  ECT completed on treadmill.
  Questionnaires:
  Total Nasal Symptom Score (TNSS 0-6). Asthma Control Test (ACT 5-25) . Positive ECT = drop in FEV1 >12% from baseline
  Interventions: Diagnostic Test: Exercise challenge test (ECT)

INTERVENTIONS:
Diagnostic Test: Exercise challenge test (ECT) — Baseline demographic, clinical and rest lung functions were recorded. ECT was performed on treadmill according to fixed protocol. Clinical data during ECT was recorded. (visit 1- performed with nose clip, visit 2- performed without nose clip). Lung function were measured and recorded at fixed time after ECT and after bronchodilator administration.

SUMMARY:
Introduction: Exercise induced bronchoconstriction (EIB) is a common finding in the pediatric population with and without asthma. EIB is suspected with a drop of 10-15% in Forced expiratory volume in the 1st second (FEV1) during exercise challenge test (ECT). Some researchers assume that oral breathing, in several mechanisms, increase hyper-responsiveness of the airways.

Aim: Asses the effect of a nose clip and allergic rhinitis in EIB. Hypothesis: The use of a nose clip in exercise challenges will increase the rate of positive tests. However, we assume that children with symptomatic allergic rhinitis will not demonstrate similar trends.

Methods: A prospective, single center cohort study in a pediatric pulmonology institute, at Ruth's children hospital, Rambam medical center, Haifa, Israel. Children referred for ECT will be registered to the study and will be evaluated in two separate visits. Visit 1 - ECT with a nose clip and visit 2 - ECT without a nose clip. Demographic and clinical data and measurements of serial vital signs, exercise data and lung functions will be taken, as well as Total Nasal Symptoms Score (TNSS) and Asthma Control Test (ACT) questionnaires.

DETAILED DESCRIPTION:
Introduction: Exercise induced bronchoconstriction (EIB) is a common finding in the pediatric population with and without asthma. EIB is evaluated with serial measurements of lung functions during exercise protocol. EIB is suspected with a drop of 10-15% in Forced expiratory volume in the 1st second (FEV1) during exercise challenge test (ECT). Some researchers assume that oral breathing, in several mechanisms, increase hyper-responsiveness of the airways.

Aim: Asses the effect of a nose clip and allergic rhinitis in exercise induced bronchoconstriction.

Hypothesis: The use of a nose clip in exercise challenges will increase the rate of positive tests. However, we assume that children with symptomatic allergic rhinitis will not demonstrate similar trends.

Methods: A prospective, single center cohort study in a pediatric pulmonology institute, at Ruth's children hospital, Rambam medical center, Haifa, Israel, during 2020-2021. Children referred for ECT will be registered to the study after signing an informed consent and will be evaluated in two separate visits. Visit 1 - ECT with a nose clip and visit 2 - ECT without a nose clip. ECT will be conducted according to the institute protocol, based on American Thoracic Society (ATS) guidelines. Demographic and clinical data and measurements of serial vital signs, exercise data and lung functions will be taken, as well as Total Nasal Symptoms Score (TNSS) and Asthma Control Test (ACT) questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Exercise challenge test as part of exercise induced asthma evaluation.
* Age 6-18 years.

Exclusion Criteria:

* Other chronic lung disease
* Significant background illness
* Severe asthma exacerbation or systemic steroids - last 2 months
* Persistent use of inhaled steroids - last 2 weeks
* Use of short acting bronchodilators - last 24 hours.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescences (6-18 years old) referred to perform exercise challenge test as a part of exercise induced asthma evaluation.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary end point | 15 minutes
  Maximum drop of forced expiratory volume in one second - (FEV1) after exercise challenge test with and without Nose clip.

SECONDARY OUTCOMES:
Secondary end point | 15 minutes
  Forced expiratory volume in one second - (FEV1) improvement after bronchodilators during exercise challenge test with and without Nose clip

CONTACTS AND LOCATIONS:
Overall Officials: Lea Bentur, MD, Principal Investigator — Rambam Medical Center Haifa, Israel.
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No